CLINICAL TRIAL: NCT04144075
Title: Application of a Mindfulness and Self-Compassion Program in Patients With Schizophrenia. Randomized Controlled Trial.
Acronym: ACAMP2020
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gutiérrez-Hernández, ME (Other)
Responsible Party: Sponsor-Investigator, Gutiérrez-Hernández, ME, Psiquiatra Adjunto. Facultativo Especialista de Área., Complejo Hospitalario Universitario Insular Materno Infantil
Organization: Complejo Hospitalario Universitario Insular Materno Infantil (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-434-1
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Schizophrenia
Keywords: Psychosis; Quality of life; Mindfulness; Compassion; Self-compassion; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mindful Self-Compassion (Experimental): Protocolized training program in mindfulness and self-compassion skills.
  Interventions: Behavioral: Mindful Self-Compassion Program
- Cognitive Behaviour Therapy Group (Active Comparator): A control intervention designed to develop a control group suitable for comparison with experimental groups receiving interventions based on mindfulness and compassion.
  Interventions: Behavioral: Cognitive Behaviour Therapy Group
- Treatment as Usual (Placebo Comparator): Es variable según las características clínicas y personales del paciente.
  Interventions: Other: Treatment as usual

INTERVENTIONS:
Behavioral: Mindful Self-Compassion Program — It is a protocolized training program in mindfulness and self-compassion skills. It has a duration of 8 weekly group sessions of about two hours and 45 minutes and a silent retreat of 4 hours.
  Other Names: CSM
  Arms: Mindful Self-Compassion
Behavioral: Cognitive Behaviour Therapy Group — It is a control intervention designed for the development of a control group suitable for comparison with experimental groups.
  Other Names: CBTG
  Arms: Cognitive Behaviour Therapy Group
Other: Treatment as usual — It is variable according to the clinical and personal characteristics of the patient, the most common components will be described.
  Other Names: TAU
  Arms: Treatment as Usual

SUMMARY:
This is a randomized clinical trial to check whether the quality of life of patients with schizophrenia improves after participation in the mindfulness and self-compassion (MSC) programme.

DETAILED DESCRIPTION:
MAIN AIM To check whether the quality of life of patients with schizophrenia improves after participation in the mindfulness and self-compassion (MSC) programme, compared with those participating in an active control programme or those following usual treatment.

DESIGN

Randomized clinical trial, three parallel groups:

1. Experimental, which will receive the MSC together with the usual treatment (TAU).
2. Active control, which will receive an alternative programme with cognitive, behavioural and psychoeducational components (CBTG) together with the TAU.
3. Passive control, which will receive the TAU. STUDY DISORDER

Schizophrenia. DATA FROM THE INTERVENTION UNDER STUDY Program developed by Kristin Neff and Christopher Germer, after observing in diverse investigations the inverse correlation between levels of self-pity and diverse pathological clinical variables.

POPULATION UNDER STUDY Patients from Telde's Mental Health Unit who have been diagnosed with schizophrenia.

TOTAL NUMBER OF SUBJECTS 150

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizohrenia

Exclusion Criteria:

* Drug addict

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-05-01 (Estimated); Primary Completion 2020-08-15 (Estimated); Study Completion 2021-02-15 (Estimated)

PRIMARY OUTCOMES:
World Health Organization Quality of Life Instument. WHOQOL-BREF | 15 minutes
  Scores from 5 to 130, the higher score the worse outcome.

SECONDARY OUTCOMES:
Self-compassion scale (SCS) | 15 minutes
  Scores from 5 to 130, the higher score the worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Díaz Megolla, Study Director — Universidad de Las Palmas de Gran Canaria